CLINICAL TRIAL: NCT03263338
Title: Mobile Health Sleep and Growth Study
Brief Title: Mobile Sleep and Growth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-014078
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Childhood Sleep Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Participants will select a time in bed target and will receive sleep tips by text messages to help reach the selected target.
  Interventions: Behavioral: Mobile Sleep and Growth Study
- Group B (Experimental): Participants will select a time in bed target and will receive sleep tips by text messages to help reach the selected target. In addition, participants in this study arm will receive additional motivational text messages beyond those given to Group A, and unique to Group B.
  Interventions: Behavioral: Mobile Sleep and Growth Study
- Group C (Experimental): Participants will select a time in bed target and will receive sleep tips by text messages to help reach the selected target. In addition, participants in this study arm will receive additional motivational text messages beyond those given to Group A, and unique to Group C.
  Interventions: Behavioral: Mobile Sleep and Growth Study

INTERVENTIONS:
Behavioral: Mobile Sleep and Growth Study — The intervention is designed to test if sleep tips delivered by text messages can aid with reaching time in bed targets. And if additional motivational text messages can further aide with reaching time in bed targets.

SUMMARY:
The purpose of this research study is to see if we can help parents to get their children to go to bed earlier. This may help children to improve their sleep. The study will use a web-based study platform and an activity monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 10 to 12 years.
2. Speak, read and write in English.
3. Parental/guardian permission (informed consent) and child assent.
4. Have a computer or a tablet computer with access to the Internet, or own a smartphone with a data and text plan.
5. Typically spend 8-9 hours in bed at night (e.g. 8 hour time in bed: go to bed at 10pm & get out of bed at 6am).

Exclusion Criteria:

1. Any clinically diagnosed sleep disorder (e.g. sleep apnea).
2. Syndromic obesity.
3. Diagnosed with a psychiatric disorder [e.g. Attention-deficit/hyperactivity disorder (ADHD), depression, anxiety].
4. Diagnosed with an eating disorder.
5. Musculoskeletal or neurological disorder that limits physical movement and activity.
6. Use of medications (prescription or otherwise) known to affect body weight and/or sleep.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Time in bed | 50-days
  Time in bed is estimated using a Fitbit activity tracker

SECONDARY OUTCOMES:
Total sleep time | 50-days
  Total sleep time is estimated using a Fitbit activity tracker

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Mitchell, Principal Investigator — Research Assistant Professor
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell JA, Morales KH, Williamson AA, Huffnagle N, Eck C, Jawahar A, Juste L, Fiks AG, Zemel BS, Dinges DF. Engineering a mobile platform to promote sleep in the pediatric primary care setting. Sleep Adv. 2021 Apr 15;2(1):zpab006. doi: 10.1093/sleepadvances/zpab006. eCollection 2021. PMID 33981997